CLINICAL TRIAL: NCT00001378
Title: A Pilot Trial of Tamoxifen and 4-HPR (4-N-Hydroxyphenyl Retinamide) in Persons at High Risk for Developing Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 940056; 94-C-0056
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-11

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: 4-Quadrant Fine Needle Aspiration; Biomarkers; Chemoprevention; Nipple Suction Aspirates; TGF Beta
MeSH Terms: conditions — Breast Neoplasms; Camurati-Engelmann Syndrome | interventions — Fenretinide

INTERVENTIONS:
Drug: fenretinide

SUMMARY:
This is a pilot, chemoprevention study. Patients receive fenretinide daily for 25 of every 28 days for 4 months and tamoxifen daily for 23 months, beginning the second month of fenretinide.

Patients are removed from study for unacceptable toxicity, the development of invasive breast cancer, or for dysfunctional uterine bleeding.

DETAILED DESCRIPTION:
This is a pilot chemo-prevention study of the combination tamoxifen and 4-HPR in persons at increased risk of developing invasive breast cancer. The objectives of the study are to determine the acute and cumulative toxicity of tamoxifen and 4-HPR in high risk persons; to assess the feasibility of obtaining adequate tissue to study potential intermediate biomarkers of proliferative disease and malignancy using nipple aspiration, four quadrant fine needle aspirates, and breast core needle biopsies; and to study the effects of tamoxifen and 4-HPR on TGF-beta isoforms and the proliferative markers ki67 and PCNA pre- and post-therapy.

ELIGIBILITY:
POPULATION CHARACTERISTICS:

Women and men at increased risk for the development of breast cancer by at least one of the following criteria:

Histologically documented ductal carcinoma in situ (DCIS), including DCIS with minimal invasion or microinvasion.

Histologically documented lobular neoplasia, including lobular hyperplasia and lobular carcinoma in situ (LCIS).

Histologically documented atypical ductal hyperplasia in postmenopausal women.

Histologically documented atypical ductal hyperplasia in premenopausal women with 1 first-degree relative (mother or sister) diagnosed with breast cancer.

Histologically documented atypical ductal hyperplasia in premenopausal women with 3 or more relatives diagnosed with breast cancer provided at least 1 is a second-degree relative.

3 or more first- or second-degree relatives diagnosed with breast or ovarian cancer with at least 1 diagnosed with breast cancer.

2 or more premenopausal (under age 50) first-degree relatives diagnosed with breast cancer.

1 or more first-degree relatives diagnosed with breast cancer if at least 1 relative in the extended pedigree had ovarian cancer.

3 or more relatives with breast cancer with at least 1 first-degree relative diagnosed with premenopausal breast cancer.

Previously diagnosed Stage I breast cancer with surgery and/or radiotherapy only (without prior adjuvant chemo- or hormonal therapy).

Positive for the BRCA1/BRCA2 gene.

No history of other invasive breast cancer.

No evidence of malignancy on breast and gynecologic exams.

Participants with a family history of breast cancer will be seen in consultation by the Family Studies Branch, NCI.

PRIOR/CONCURRENT THERAPY:

Mastectomy or lumpectomy plus radiotherapy required prior to entry for patients with DCIS. Patients with DCIS who have participated in protocol NCI-MB-348 eligible.

No participation in any other breast cancer prevention study involving pharmacologic intervention.

No prior chemotherapy or hormonal therapy for invasive breast cancer.

At least 3 months since estrogen or progesterone replacement therapy or hormonal contraceptives.

PATIENT CHARACTERISTICS:

Age: 35 and over.

Performance status: Ambulatory.

Life expectancy: At least 10 years.

Hematopoietic: Complete blood count normal.

Hepatic:

Bilirubin normal.

Alkaline phosphate normal.

AST normal.

PT, PTT normal.

No history of bleeding disorder.

No history of chronic hepatitis or cirrhosis.

Renal:Creatinine less than 1.5 mg/dL.

Cardiovascular:

No history of deep venous thrombosis.

No history of pulmonary embolus.

Other:

No allergy to any study medication.

Capable of tolerating multiple diagnostic procedures.

No history of abnormal vaginal bleeding. Hysterectomy for vaginal bleeding of benign etiology allowed.

No history of retinal disease, macular degeneration, or night blindness.

No medical or psychiatric risk due to nonmalignant systemic disease that would preclude study participation.

No history of malignancy except: Curatively treated nonmelanomatous skin cancer. Curatively treated in situ cervical carcinoma. Hodgkin's disease treated more than 5 years ago.

No pregnant women.

Adequate contraception required of fertile patients during and for 12 months after fenretinide and for 2 months after tamoxifen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 1994-01; Study Completion 2000-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] London SJ, Connolly JL, Schnitt SJ, Colditz GA. A prospective study of benign breast disease and the risk of breast cancer. JAMA. 1992 Feb 19;267(7):941-4. PMID 1734106
- [Background] Dupont WD, Page DL. Risk factors for breast cancer in women with proliferative breast disease. N Engl J Med. 1985 Jan 17;312(3):146-51. doi: 10.1056/NEJM198501173120303. PMID 3965932